CLINICAL TRIAL: NCT03880435
Title: The Cost-effectiveness of Anti-adhesion Treatment With HYALOBARRIER® GEL ENDO Versus no Gel Following the Removal by Hysteroscopy of Endometrial Polyps, Fibroids With Uterine Cavity Deformation, Uterine Septa, Intrauterine Adhesions or Retained Products of Conception for Improving Reproductive Outcome in Women Wishing to Become Pregnant: a Multi-centre, Parallel Group, Superiority, Double-blind, Randomized Controlled Trial
Brief Title: HYALOBARRIER® GEL ENDO Versus no HYALOBARRIER® GEL ENDO Following Operative Hysteroscopy for Improving Reproductive Outcome in Women With Intrauterine Pathology Wishing to Become Pregnant
Acronym: AGNOHSTIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government); Nordic Pharma SAS (Industry); Universitaire Ziekenhuizen KU Leuven (Other); Universitair Ziekenhuis Brussel (Other); Health, Innovation and Research Institute (HIRUZ) UZ Ghent (Unknown); University of Liege (Other); UCL Bruxelles (Unknown); Jessa hospital, Hasselt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AGNOHSTIC
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Infertility; Polyp Uterus; Myoma;Uterus; Adhesion; Hysteroscopy; Uterine Septum; Retained Products of Conception
Keywords: Infertility; Reproductive outcome; Hysteroscopy; Adhesion prophylaxis
MeSH Terms: conditions — Infertility; Myofibroma; Tissue Adhesions; Septate Uterus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: None of the participants will be informed of the allocated treatment by the surgeon performing the operative hysteroscopy or the personnel present in the OR. The medical record will not reveal any information whether HYALOBARRIER® GEL ENDO was applied at the end of the procedure. The REDCap software will automatically document the allocation and store all the records and the randomisations. The gynaecologist doing the operative hysteroscopy should not be the same as the fertility physician and the gynaecologist doing the second look hysteroscopy. In the exceptional case that the surgeon doing the operative hysteroscopy is the same person as the fertility physician or the gynaecologist doing the second-look hysteroscopy, blinding is assured by notification of treatment allocation if the surgeon has left the operating room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyalobarrier® gel endo (Experimental): Application of Hyalobarrier® gel endo immediate after the complete hysteroscopic removal of the polyp, myoma, adhesion, uterine septum or retained products of conception + application of sterile ultrasound gel into the vagina (to blind all trial participants, fertility physicians and gynaecologists doing second-look hysteroscopy)
  Interventions: Device: Hyalobarrier® gel endo
- No Hyalobarrier® gel endo (No Intervention): No application of Hyalobarrier® gel endo after the hysteroscopic removal of the polyp, myoma, adhesion, uterine septum or retained products of conception + application of sterile ultrasound gel into the vagina (to blind all trial participants, fertility physicians and gynaecologists doing second- or third-look hysteroscopy)

INTERVENTIONS:
Device: Hyalobarrier® gel endo — Intra-uterine application of 10ml sterile gel containing 30mg APC. It will be administered once, peroperatively immediate after the complete hysteroscopic removal of the polyp, myoma, adhesion, uterine septum or retained products of conception
  Arms: Hyalobarrier® gel endo

SUMMARY:
To compare the costs and effects of HYALOBARRIER® GEL ENDO versus no HYALOBARRIER® GEL ENDO for increasing the chance of conception leading to live birth measured at 30 weeks after randomization in women wishing to become pregnant after surgical removal of intrauterine pathology (endometrial polyps, fibroids with uterine cavity deformation, uterine septa, IUAs or RPOC after miscarriage) by hysteroscopy as an outpatient or in hospital treatment.

DETAILED DESCRIPTION:
Design:

Multi-centre, parallel group, superiority, double-blind, randomized controlled trial. Post market study of a Medical Device class III.

Participant:

Women aged 18 to 47 years attending Belgian gynaecological departments, scheduled for operative hysteroscopy for endometrial polyps, fibroids with uterine cavity deformation, uterine septa, intrauterine adhesions (IUAs) or retained products of conception, and wishing to conceive spontaneously or before fertility treatment with ovulation induction (OI), controlled ovarian stimulation (COS), intrauterine insemination (IUI) or IVF/ICSI.

Treatment:

Application of Hyalobarrier® gel endo at time of surgery

Control:

No application of Hyalobarrier® gel endo

Follow up:

short term follow-up: 30 weeks after receiving the treatment allocation long term follow-up: 66 weeks after receiving the treatment allocation

To blind all trial participants, fertility physicians and gynaecologists doing second- or third-look hysteroscopy, 10 ml of a sterile ultrasound gel will be applied into the vagina at the end of the procedure in all women regardless of their treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18 to 47 years attending Belgian fertility clinics, scheduled for operative hysteroscopy for endometrial polyps, fibroids with uterine cavity deformation, uterine septa, intrauterine adhesions (IUAs) and retained products of conception, and wishing to conceive spontaneously or before fertility treatment with ovulation induction (OI), controlled ovarian stimulation (COS), intrauterine insemination (IUI) or IVF/ICSI.

Exclusion Criteria:

* Women younger than 18 years
* Women 48 years of age or older
* Women with a known allergy to HYALOBARRIER® GEL ENDO
* Women with an active infection of the genital tract proven by genital swabs for PCR (Chlamydia, gonococci) or endometrial biopsy (endometritis), not treated at the time of the pre- screening visit. Women adequately treated with proven cure (negative swabs or normal endometrial biopsy) can be included
* Subserosal fibroids (FIGO or PALM-COEIN classification type 6, 7) - leiomyomas that originate from the myometrium at the serosa of the uterus or intramural fibroids without uterine cavity deformation as documented by ultrasound, hysterography or hysteroscopy - as the sole uterine cavity abnormality identified in the screening phase.
* Women with fibroids, polyps, uterine septa or IUAs suffering from other symptoms, for instance abnormal uterine bleeding, but not wishing to conceive from 6 weeks following surgery
* Women with other Müllerian tract anomalies other than a uterine septum as the sole uterine cavity abnormality identified in the screening phase
* Women who participated in the trial but failed to conceive and who present with a recurrence of polyps, fibroids with cavity deformation, uterine septum or IUAs
* Women who refuse to give written informed consent.

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 419 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Conception leading to live birth | > 30 weeks after randomisation
  the amount of clinical pregnancies at 30 weeks after randomisation, leading to live birth (at least one live foetus after 20 weeks of gestation, that resulted in at least one live baby (the investigators counted the delivery of singleton, twin or multiple pregnancies as one live birth)

SECONDARY OUTCOMES:
Time to conception | < 30 weeks after receiving treatment allocation
  the time from receiving the allocated treatment to the date of conception
Clinical pregnancy | < 30 weeks after receiving treatment allocation
  An ultrasound visible gestational sac
Miscarriage | < 30 weeks after receiving treatment allocation
  a spontaneous loss of pregnancy before 20 completed weeks of gestational age, or if gestational age is unknown, the loss of an embryo/fetus of less than 400 grams
Ectopic pregnancy | < 30 weeks after receiving treatment allocation
  a pregnancy in which implantation takes place outside the uterine cavity
Adhesions | > 30w after receiving treatment allocation (in women who failed to conceive)
  The severity will be scored according to the revised American Fertility Society (AFS) scoring system
Pre-eclampsia | > 30 weeks after receiving treatment allocation
  Pre-eclampsia in women who conceived during the study period, leading to an ongoing pregnancy beyond 20 weeks of gestation
Preterm birth | > 30 weeks after receiving treatment allocation
  Preterm birth in women who conceived during the study period, leading to an ongoing pregnancy beyond 20 weeks of gestation
Stilbirth | > 30 weeks after receiving treatment allocation
  Stillbirth in women who conceived during the study period, leading to an ongoing pregnancy beyond 20 weeks of gestation
Low/very low birth weight (gram) | > 30 weeks after receiving treatment allocation
  low/very low birth weight (gram) in women who conceived during the study period, leading to an ongoing pregnancy beyond 20 weeks of gestation
Caesarean section rates | > 30 weeks after receiving treatment allocation
  caesarean section rates in women who conceived during the study period, leading to an ongoing pregnancy beyond 20 weeks of gestation
Neonatal complications | > 30 weeks after receiving treatment allocation
  Neonatal complications in women who conceived during the study period,
The total hospital bill | measured at the time of diagnosis of an ongoing pregnancy by the detection at 12 weeks in a clinical pregnancy of a positive heart beat on ultrasound examination
  Direct health-related costs

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weyers, MD,PhD, Principal Investigator — Women's Clinic
Locations (1):
- University hospital Ghent, Ghent, East-Flanders, Belgium

REFERENCES:
- [Background] Acunzo G, Guida M, Pellicano M, Tommaselli GA, Di Spiezio Sardo A, Bifulco G, Cirillo D, Taylor A, Nappi C. Effectiveness of auto-cross-linked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic adhesiolysis: a prospective, randomized, controlled study. Hum Reprod. 2003 Sep;18(9):1918-21. doi: 10.1093/humrep/deg368. PMID 12923149
- [Background] Bosteels J, Weyers S, Kasius J, Broekmans FJ, Mol BW, D'Hooghe TM. Anti-adhesion therapy following operative hysteroscopy for treatment of female subfertility. Cochrane Database Syst Rev. 2015 Nov 9;(11):CD011110. doi: 10.1002/14651858.CD011110.pub2. PMID 26559098
- [Background] Casini ML, Rossi F, Agostini R, Unfer V. Effects of the position of fibroids on fertility. Gynecol Endocrinol. 2006 Feb;22(2):106-9. doi: 10.1080/09513590600604673. PMID 16603437
- [Background] Di Spiezio Sardo A, Spinelli M, Bramante S, Scognamiglio M, Greco E, Guida M, Cela V, Nappi C. Efficacy of a polyethylene oxide-sodium carboxymethylcellulose gel in prevention of intrauterine adhesions after hysteroscopic surgery. J Minim Invasive Gynecol. 2011 Jul-Aug;18(4):462-9. doi: 10.1016/j.jmig.2011.04.007. PMID 21777835
- [Background] Farhi J, Orvieto R. Cumulative clinical pregnancy rates after COH and IUI in subfertile couples. Gynecol Endocrinol. 2010 Jul;26(7):500-4. doi: 10.3109/09513590903367036. PMID 20540664
- [Background] Farquhar C, Lilford RJ, Marjoribanks J, Vandekerckhove P. Laparoscopic 'drilling' by diathermy or laser for ovulation induction in anovulatory polycystic ovary syndrome. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD001122. doi: 10.1002/14651858.CD001122.pub3. PMID 17636653
- [Background] Gnoth C, Godehardt D, Godehardt E, Frank-Herrmann P, Freundl G. Time to pregnancy: results of the German prospective study and impact on the management of infertility. Hum Reprod. 2003 Sep;18(9):1959-66. doi: 10.1093/humrep/deg366. PMID 12923157
- [Background] Guida M, Acunzo G, Di Spiezio Sardo A, Bifulco G, Piccoli R, Pellicano M, Cerrota G, Cirillo D, Nappi C. Effectiveness of auto-crosslinked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic surgery: a prospective, randomized, controlled study. Hum Reprod. 2004 Jun;19(6):1461-4. doi: 10.1093/humrep/deh238. Epub 2004 Apr 22. PMID 15105384
- [Background] Jansen FW, Vredevoogd CB, van Ulzen K, Hermans J, Trimbos JB, Trimbos-Kemper TC. Complications of hysteroscopy: a prospective, multicenter study. Obstet Gynecol. 2000 Aug;96(2):266-70. doi: 10.1016/s0029-7844(00)00865-6. PMID 10908775
- [Background] Kasius JC, Broekmans FJ, Veersema S, Eijkemans MJ, van Santbrink EJ, Devroey P, Fauser BC, Fatemi HM. Observer agreement in the evaluation of the uterine cavity by hysteroscopy prior to in vitro fertilization. Hum Reprod. 2011 Apr;26(4):801-7. doi: 10.1093/humrep/der003. Epub 2011 Feb 9. PMID 21310749
- [Background] McLernon DJ, Maheshwari A, Lee AJ, Bhattacharya S. Cumulative live birth rates after one or more complete cycles of IVF: a population-based study of linked cycle data from 178,898 women. Hum Reprod. 2016 Mar;31(3):572-81. doi: 10.1093/humrep/dev336. Epub 2016 Jan 18. PMID 26783243
- [Background] Perez-Medina T, Bajo-Arenas J, Salazar F, Redondo T, Sanfrutos L, Alvarez P, Engels V. Endometrial polyps and their implication in the pregnancy rates of patients undergoing intrauterine insemination: a prospective, randomized study. Hum Reprod. 2005 Jun;20(6):1632-5. doi: 10.1093/humrep/deh822. Epub 2005 Mar 10. PMID 15760959